CLINICAL TRIAL: NCT01731067
Title: Cocktail Approach for Cytochrome P450 and P-glycoprotein Activity Assessment Using Dried Blood Spot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jules Desmeules (Other)
Responsible Party: Sponsor-Investigator, Jules Desmeules, Pr, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Coktail DBS
Record Dates: First submitted 2012-11-14; First posted 2012-11-21 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Bupropion; Flurbiprofen; Omeprazole; Dextromethorphan; Midazolam; fexofenadine; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CYP1A2, 2B6, 2C9, 2C19, 3A4 inhibitors (Active Comparator): Oral intake of fluvoxamine (50 mg per day during 2 days) and voriconazole (400 mg) before oral intake of the cocktail probe drugs
  Interventions: Drug: Cocktail probe drugs
- CYP2D6 and P-gp inhibitor (Active Comparator): Oral intake of quinidine (200 mg) before oral intake of the cocktail probe drugs
  Interventions: Drug: Cocktail probe drugs
- CYPs and P-gp inducer (Active Comparator): Oral intake of rifampicin (600 mg per day during 7 days) before oral intake of the cocktail probe drugs
  Interventions: Drug: Cocktail probe drugs
- Probe cocktail alone (Experimental): Oral intake of the cocktail probe drugs :
  * bupropion 25 mg
  * flurbiprofen 25 mg
  * omeprazole 5 mg
  * dextromethorphan 5 mg
  * midazolam 1 mg
  * fexofenadine 25mg
  * Caffeine (a cup of coffee)
  Interventions: Drug: Cocktail probe drugs

INTERVENTIONS:
Drug: Cocktail probe drugs
  Other Names: Oral intake of the cocktail probe drugs :; bupropion 25 mg; flurbiprofen 25 mg; omeprazole 5 mg; dextromethorphan 5 mg; midazolam 1 mg; fexofenadine 25mg; Caffeine (a cup of coffee)

SUMMARY:
Phenotyping is an approach largely used for the evaluation of the activity of cytochromes and transporters in vivo. It consists of the administration of probe substances metabolised by a specific cytochrome or transported by P-glycoprotein (P-gp) for example, followed by the determination of a metabolic ratio or the evaluation of the plasmatic or urinary concentrations of the probe substances. The administration of a cocktail containing several probe substances allows the simultaneous evaluation of the activity of several cytochromes and P-gp in a single test.

The aim of this project is the validation of a phenotyping cocktail of low dose probe drugs for the assessment of cytochrome P450 and P-gp activities by simple capillary blood sampling and dried blood spot (DBS) analysis. The cocktail consists of caffeine, bupropion, flurbiprofen, omeprazole, dextromethorphan, midazolam and fexofenadine for the simultaneous phenotyping of CYP1A2, CYP2B6, CYP2C9, CAP2C19, CYP2D6, CYP3A4 and P-gp, respectively.

The modulation of the activity of cytochromes or P-gp will be evaluated by the administration of inhibitors (fluvoxamine, voriconazole, quinidine) or inducer (rifampicin) of the metabolic pathways or the P-gp mediated transport.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged from 18 to 60 years
* BMI between 18 and 25
* Understanding of French language and able to give a written inform consent.

Exclusion Criteria:

* Smoker
* Taking drugs which alter CYPs activity
* Renal or hepatic impairment
* Medical history of porphyria
* Medical history of chronic alcoholism or abuse of psychoactive drugs
* Liver transplantation
* Sensitivity to any of the drugs used
* Wearing contact lenses (risk of coloration with rifampicin)
* ECG showing long QT interval (>0.46sec)
* Alteration of hepatic tests
* Presenting genetic polymorphism of poor CYP 2B6, 2C9, 2C19, 2D6 metabolisers

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Probe cocktail drugs plasma and capillary concentrations in presence/absence of CYP1A2,2B6, 2C9, 2C19, 2D6, 3A4 and P-gp inhibitor or inducer | 4 singles days spaced out with one week wash-out periods

SECONDARY OUTCOMES:
correlation between plasma or urine and capillary concentrations for each probe cocktail drug | 4 singles days spaced out with one week wash-out periods
comparison. between genotype and phenotype for each enzyme | one day

CONTACTS AND LOCATIONS:
Overall Officials: Jules A Desmeules, Pr, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Bosilkovska M, Samer CF, Deglon J, Rebsamen M, Staub C, Dayer P, Walder B, Desmeules JA, Daali Y. Geneva cocktail for cytochrome p450 and P-glycoprotein activity assessment using dried blood spots. Clin Pharmacol Ther. 2014 Sep;96(3):349-59. doi: 10.1038/clpt.2014.83. Epub 2014 Apr 10. PMID 24722393